CLINICAL TRIAL: NCT01928238
Title: Physiologic Effects of Noninvasive Neurally Adjusted Ventilatory Assist (NAVA) Versus Noninvasive Pressure Support Ventilation in Patients at Risk for Respiratory Distress Needed Preventive Used of Noninvasive Ventilation After Extubation.
Acronym: NAVA-VNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2011/27
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-01

CONDITIONS: Acute Respiratory Distress
Keywords: NIV; NAVA; noninvasive neurally adjusted ventilatory; noninvasive pressure support ventilation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Patients will have two 20-minute noninvasive periods :
  Noninvasive neurally adjusted ventilatory assist (NIV-NAVA) and then Noninvasive pressure support ventilation (NPSV)
  Interventions: Device: Noninvasive neurally adjusted ventilatory assist (NIV-NAVA).; Device: Noninvasive pressure support ventilation (NPSV)
- Arm 2 (Experimental): Patients will have two 20-minute noninvasive periods :
  Noninvasive pressure support ventilation (NPSV) and then Noninvasive neurally adjusted ventilatory assist (NIV-NAVA)
  Interventions: Device: Noninvasive neurally adjusted ventilatory assist (NIV-NAVA).; Device: Noninvasive pressure support ventilation (NPSV)

INTERVENTIONS:
Device: Noninvasive neurally adjusted ventilatory assist (NIV-NAVA).
Device: Noninvasive pressure support ventilation (NPSV)

SUMMARY:
The purpose of this study is to compare inspiratory effort, comfort, gas exchange and patient ventilator synchrony during non-invasive neurally adjusted ventilatory assist or pneumatically triggered and cycled-off noninvasive pressure support ventilation (NPSV), in patient at risk of respiratory distress after extubation.

DETAILED DESCRIPTION:
Reintubation, which occurs after planned extubation, is a relevant consequence of respiratory failure after extubation. The early use of noninvasive pressure support ventilation averted respiratory failure after extubation in patients at increased risk. However patient tolerance to the technique is a critical factor determining its success. One of the key factors determining tolerance to Non Invasive Ventilation (NIV) is optimal synchrony between the patient's spontaneous breathing activity and the ventilator's settings, known as patient ventilator interaction. Optimal patient-ventilator synchrony during NIV can prove very difficult to achieve due to the presence of leaks, the type of interface which can interfere with various aspects of ventilator function. Patient ventilator synchrony during NPSV can be compromised when using conventional pneumatic triggering, with the ventilator-delivered inspiratory support starting after the patient's inspiratory effort. The switch from inspiration to expiration (cycling-off) should, ideally, coincide with the end of the patient's inspiratory effort. However greater asynchrony at the end of inspiration, with the ventilator cycling off either too early or too late compared to the end of the patient's inspiratory effort can be observed during NPSV. A possible solution is to replace the pneumatic triggering with neural triggering and cycling off using the diaphragm electrical activity (Eadi). Neurally adjusted ventilatory assist (NAVA) uses the electrical activity of the diaphragm to control the timing and pressure of the ventilation delivered. The ventilator is triggered, limited and cycled-off directly by Eadi. The Eadi is measured by a multiple array oesophageal electrode. The array of bipolar electrodes can be mounted on a feeding tube, which is routinely introduced in critically ill patients.

ELIGIBILITY:
inclusion criteria:

* Patients intubated for 48 h or more
* Patients who tolerated a 120-min spontaneous breathing trial after recovery from their acute disease with no signs of respiratory failure
* Patients at high risk for respiratory after extubation were enrolled if they had at least two of the following risk factors for respiratory failure after extubation:

  * age older than 65 years
  * Chronic obstructive pulmonary disease,
  * heart failure as the cause for intubation
  * An Acute Physiology and Chronic Health Evaluation (APACHE)-II score greater than 12 on the day of extubation.

exclusion criteria:

* Age younger than 18 years
* Head trauma or surgery
* Recent gastric or oesophageal surgery
* Active upper gastrointestinal bleeding
* Excessive amount of respiratory secretions
* Poor cooperation
* Decision to limit life-supporting treatments in the ICU
* Tracheostomy or other upper airway disorders
* Lack of collaboration
* Do not resuscitate order or any decision to limit therapeutic effort in the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle effort | At inclusion (day 0)
  The primary endpoint variable is the inspiratory muscle effort. To estimate the inspiratory effort, we will determine the transdiaphragmatic pressure (Pdi), the transdiaphragmatic pressure time product per breath (PTPdi/b) or per minute (PTPdi/min) and the Electrical Activity of the Diaphragm (EADI)max.

SECONDARY OUTCOMES:
patient ventilator synchrony | At inclusion (Day 0)
  Patient ventilator synchrony will be identified by estimating the following variables: autocycled breaths, ineffective inspiratory effort, the inspiratory trigger delay, the expiratory trigger delay and the time of synchrony between muscle effort and ventilator support.
gas exchange | At inclusion (Day 0)
Patient comfort | At inclusion (Day 0)
  Patient comfort will be assessed using a five-item semi quantitative scale: 1, uncomfortable; 2, somewhat uncomfortable; 3, acceptable; 4, somewhat comfortable; and 5, comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VARGAS, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France